CLINICAL TRIAL: NCT04959838
Title: Monitoring of JOB STRESS Related to Night Shifts in OPHthalmology Physicians and Residents
Brief Title: JOB STRESS in OPHthalmology Physicians and Residents
Acronym: JOBSTRESS-OPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Clermont Auvergne (UCA), Clermont-Ferrand, France (Unknown); LaPSCO laboratory, UMR CNRS 6024, Clermont-Ferrand, France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RBHP 2020 DUTHEIL 2; 2020-A03231-38 (Other: 2020-A03231-38)
Record Dates: First submitted 2021-06-22; First posted 2021-07-13 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Stress; Heart Rate Variability
Keywords: ophthalmologists; on-call duty; stress; surgical simulator; heart rate variability; sleep; questionnaires; actimetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ophthalmology physicians and residents (Experimental): Ophthalmology physicians and residents will be followed during 34h, from 8 am to 6 pm the following day,in five different conditions:
  * Control day (no work)
  * Typical working day
  * Working day + one night shift
  * Emergency working day + two consecutive night shifts
  * Night shift.
  Interventions: Behavioral: Impact of prolonged work

INTERVENTIONS:
Behavioral: Impact of prolonged work — Evaluate the impact of prolonged work (up to 60 consecutive hours) on the surgical capacities evaluated on a simulator, as well as on stress markers (questionnaires, saliva assays, skin conductance, quality of sleep) compared to a standard day.

SUMMARY:
Ophthalmology physicians and residents work under stress conditions during night emergency ophthalmology shifts. Under time pressure, that is a characteristic of the urgency of care, they must use all their cognitive resources to make an accurate diagnosis and to provide accurate decisions, with sometimes surgical emergency acts. In addition, in France, they work at night following by an usual day work, and they can also work 48 consecutive hours during weekends, followed by a work day … i.e. 60 consecutive hours of work … Long working hours with a short recovery time has been demonstrated to be a major factor of stress and fatigue. Even if not demonstrated on ophthalmologists, those working conditions may contribute to symptoms of mental exhaustion and physical fatigue (sleep deprivation), often accompanied by a loss of motivation at work. This may leads to a feeling of loss of time control; stress can also distort the perception of time and leads to hasty actions or delayed decision-making. The combined effects of stress, feelings of loss of time control, and fatigue necessarily have an impact on work performance and work quality, with a high risk of medical error. Moreover, prolonged stress may expose ophthalmologists to a higher risk of multiple diseases, predominantly systemic inflammation and coronary heart disease.

The main hypothesis is that prolonged work (up to 60 consecutive working hours) may impact on HRV, comparatively to a typical working day.

DETAILED DESCRIPTION:
The JOBSTRESS.OPH protocol was designed to study the impact of prolonged work (up to 60 consecutive working hours) on HRV, comparatively to a typical working day. Each residents and / or ophthalmology physicians participates up to a maximum of 5 times. Participants wears a heart rate belt and a watch that measures physical activity and skin conductance for 34 hours straight. Participants only wears an EEG monitor while sleeping to assess its quality. At the end of the evaluation session, a simulator test mimicking the successive stages of cataract surgery is performed, as well as the performance of saliva tests. Short quality of life assessment questionnaires are completed at the start and end of the day, supplemented by a general questionnaire completed only once during the study.

Statistical analysis will be performed using Stata software (v15, Stata-Corp, College Station, US). Categorical parameters will be described in terms of numbers and frequencies, whereas continuous variables will be expressed as mean and standard deviation or median and [inter-quartile range] according to statistical distribution. All statistical tests will be two-sided and p<0.05 will be considered significant. Graphic representations will be complete presentations of results.

Investigators process multivariate physiological series (HRV, SC, biomarkers) in order to build a stress index. For such multivariate physiological series, investigators first use change point analysis on each univariate series in order to get clusters with constant parameters, then investigators use classification algorithm on the constant parameters obtained in first step in order to obtain different classes corresponding to different levels of stress. Eventually, investigators obtain at each time the level of stress and can compare it to the environmental conditions.

ELIGIBILITY:
Inclusion Criteria:

* Ophthalmologists defined as physicians who completed the ophthalmology DES (Specialized studies diploma), as well as ophthalmology residents defined as a resident registered in the ophthalmology DES working during the inclusion period in the ophthalmology department of the university hospital center of Clermont-Ferrand.
* Ability to give a written informed consent to participate in research.
* Affiliation to a social security system.
* Age between 18 and 65 years old

Exclusion Criteria:

* Participant refusal to participate
* Children under the age of 18, pregnant and breastfeeding women, protected adults (individuals under guardianship by court order), adults deprived of their liberty.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | During 34 hours in the five different conditions
  HRV will be explored in time and frequency domains Abrupt changes in HRV signals will be explored.

SECONDARY OUTCOMES:
change in stress levels | at 8am, beginning of the 34 hours follow-up, in the five different conditions
  measure of stress using visual analogue scale of 100 mm, from 0 to 100. Higher scores mean a worse outcome level.
change in stress levels | at 6pm, end of the 34 hours follow-up, in the five different conditions
  measure of stress using visual analogue scale of 100 mm, from 0 to 100. Higher scores mean a worse outcome level.
change in fatigue levels | at 8am, beginning of the 34 hours follow-up, in the five different conditions
  measure of fatigue using visual analogue scale of 100 mm, from 0 to 100. Higher scores mean a worse outcome level.
change in fatigue levels | at 6pm, end of the 34 hours follow-up, in the five different conditions
  measure of fatigue using visual analogue scale of 100 mm, from 0 to 100. Higher scores mean a worse outcome level.
change in burnout levels | at 8am, beginning of the 34 hours follow-up, in the five different conditions
  measure of burnout using visual analogue scale of 100 mm, from 0 to 100. Higher scores mean a worse outcome level.
change in burnout levels | at 6pm, end of the 34 hours follow-up, in the five different conditions
  measure of burnout using visual analogue scale of 100 mm, from 0 to 100. Higher scores mean a worse outcome level.
change in depression levels | at 8am, beginning of the 34 hours follow-up, in the five different conditions
  measure of depression using visual analogue scale of 100 mm, from 0 to 100. Higher scores mean a worse outcome level.
change in depression levels | at 6pm, end of the 34 hours follow-up, in the five different conditions
  measure of depression using visual analogue scale of 100 mm, from 0 to 100. Higher scores mean a worse outcome level.
change in anxiety levels | at 8am, beginning of the 34 hours follow-up, in the five different conditions
  measure of anxiety using visual analogue scale of 100 mm, from 0 to 100. Higher scores mean a worse outcome level.
change in anxiety levels | at 6pm, end of the 34 hours follow-up, in the five different conditions
  measure of anxiety using visual analogue scale of 100 mm, from 0 to 100. Higher scores mean a worse outcome level.
change in "Job demand control support" levels | at 8am, beginning of the 34 hours follow-up, in the five different conditions
  measure of job demand, job control and support levels using visual analogue scale of 100 mm, from 0 to 100. Higher scores of demand mean a worse level. Higher scores of control and support mean a better level.
change in "Job demand control support" levels | at 6pm, end of the 34 hours follow-up, in the five different conditions
  measure of job demand, job control and support levels using visual analogue scale of 100 mm, from 0 to 100. Higher scores of demand mean a worse level. Higher scores of control and support mean a better level.
change in "Effort reward imbalance" levels | at 8am, beginning of the 34 hours follow-up, in the five different conditions
  measure of effort reward imbalance using visual analogue scale of 100 mm, from 0 to 100. Higher scores of mean a better outcome level.
change in "Effort reward imbalance" levels | at 6pm, end of the 34 hours follow-up, in the five different conditions
  measure of effort reward imbalance using visual analogue scale of 100 mm, from 0 to 100. Higher scores of mean a better outcome level.
change in work addiction levels | at 8am, beginning of the 34 hours follow-up, in the five different conditions
  measure of work addiction using visual analogue scale of 100 mm, from 0 to 100. Higher scores mean a worse outcome level.
change in work addiction levels | at 6pm, end of the 34 hours follow-up, in the five different conditions
  measure of work addiction using visual analogue scale of 100 mm, from 0 to 100. Higher scores mean a worse outcome level.
change in sleep quality | at 8am, beginning of the 34 hours follow-up, in the five different conditions
  measure of sleep quality using visual analogue scale of 100 mm, from 0 to 100. Higher scores mean a worse outcome level.
change in sleep quality | at 6pm, end of the 34 hours follow-up, in the five different conditions
  measure of sleep quality using visual analogue scale of 100 mm, from 0 to 100. Higher scores mean a worse outcome level.
Saliva biomarkers cortisol | baseline of the 34 hours procedure, in the five different conditions
  measure on Cortisol
Saliva biomarkers cortisol | 24hours after the beginning of the procedure, in the five different conditions
  measure on Cortisol
Saliva biomarkers dheas | baseline of the 34 hours procedure, in the five different conditions
  measure on dheas
Saliva biomarkers dheas | 24 hours after the beginning of the procedure, in the five different conditions
  measure on dheas
Saliva biomarkers lgAs | baseline of the 34 hours procedure, in the five different conditions
  measure on lgAs
Saliva biomarkers lgAs | 24 hours after the beginning of the procedure, in the five different conditions
  measure on lgAs
Saliva biomarkers Leptine | baseline of the 34 hours procedure, in the five different conditions
  measure on Leptine
Saliva biomarkers Leptine | 24 hours after the beginning of the procedure, in the five different conditions
  measure on Leptine
Saliva biomarkers Ghrelin | baseline of the 34 hours procedure, in the five different conditions
  measure on Ghrelin
Saliva biomarkers Ghrelin | 24 hours after the beginning of the procedure, in the five different conditions
  measure on Ghrelin
Declared level of physical activity | once at 8am, at the beginning of the procedure
  Physical activity is assessed with one question
Level of physical activity | during 34 hours, in the five different conditions
  Physical activity is assessed with a 3-Axis accelerometer
Level of sedentary | once at 8am, at the beginning of the procedure
  Sedentary is assessed regarding the time spent sitting assessed with one question
Food intake | 34 hours recording, in the five different conditions
  assessing food intake with ingesta
Sick leave | once at 8am, at the beginning of the procedure
  assessing the number of absence days the previous 6 months using a questionnaire
Height | once at 8am, at the beginning of the procedure
  measure of height in cm using a questionnaire
Weight | once at 8am, at the beginning of the procedure
  measure of weight in kilograms using a questionnaire
Age | once at 8am, at the beginning of the procedure
  measure of age in years using a questionnaire
Gender | once at 8am, at the beginning of the procedure
  measure of gender using a questionnaire
Qualification | once at 8am, at the beginning of the procedure
  measure of qualification using a questionnaire
Personal status | once at 8amat the beginning of the procedure
  measure of personal status using a questionnaire
Lifestyle | once at 8am, at the beginning of the procedure
  Assessing factors related to lifestyle as smoking, alcohol and coffee consumption using a questionnaire
Skin conductance | during 34 hours , in the five different conditions
  measure of the skin conductance using Wrist band electrodes
Sleep quality | measure for about 7 hours the night of the control day (no work)
  measure of sleep quality using Sleep profiler
Sleep quality | measure for about 7 hours during the night of the typical working day
  measure of sleep quality using Sleep profiler
Surgical performance | Once at 6pm, at the end of the 34 hours follow-up , in the five different conditions
  assessing surgical performance using a high-end virtual reality simulator for intraocular surgery training

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric DUTHEIL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France